CLINICAL TRIAL: NCT03586947
Title: Association Between Vitamin D and the Risk of Uterine Fibroids
Acronym: ABVDATROUF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2017-07-101
Record Dates: First submitted 2018-06-12; First posted 2018-07-16 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-07

CONDITIONS: Gynaecological Disease; Vitamin D Deficiency; Uterine Fibroids
MeSH Terms: conditions — Genital Diseases, Female; Vitamin D Deficiency; Leiomyoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D3 Drops group (Experimental): Patients in this group would take Vitamin D3 400 UNT Oral Capsule.
  Interventions: Drug: Vitamin D3 400 UNT Oral Capsule
- Non-Vitamin D3 Drops group (No Intervention): Patients in this group would take nothing.

INTERVENTIONS:
Drug: Vitamin D3 400 UNT Oral Capsule — 50,000 IU of vitamin D once a week for 8 weeks, 1500-2000 IU/day.
  Other Names: Vitamin D3 drops
  Arms: Vitamin D3 Drops group

SUMMARY:
The aim of this randomised clinical trial study is to evaluate whether supplementation with vitamin D could reduce the risk of uterine fibroids in reproductive stage women.

DETAILED DESCRIPTION:
A total of 1160 hypovitaminosis D patients (12 ng/ml ≤ serum 25-hydroxyvitamin D3 < 20 ng/ml) without uterine fibroids will be randomly assigned in a ratio of 1:1 to two groups: intervention group and control group. The intervention group will receive 1600 IU/d of vitamin D3; the control group will receive regular follow-up. Patients will be followed up at the same time points for 24 months. The outcome measure is the incidence of uterine fibroids in different groups.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the study with informed consent;
2. Females aged 35-50 who are confirmed with a normal, fibroid-free uterine structure, by means of transvaginal or abdominal ultrasonography;
3. Serum25-hydroxyvitamin D3 <20 ng/ml, ≥ 12ng/ml.

Exclusion Criteria:

1. Use of sexual hormone, mifepristone, gonadotropin-releasing hormone agonist (GnRHa), or other medication which is likely to interfere with uterine fibroids within 3 months;
2. Pregnancy, lactation, postmenopause, or planned pregnancy within two years;
3. Allergic to vitamin D3;
4. Suspected or identified as other tumors of genital tract;
5. History of hysterectomy or myomectomy;
6. History of osteoporosis or vitamin D deficiency taking vitamin D supplements within previous one month;
7. History of hyperparathyroidism, infectious diseases (tuberculosis, AIDS), autoimmune diseases, or digestive system diseases (malabsorption, crohn disease and dysentery);
8. Alanine aminotransferase (ALT) or aspartate transaminase (AST) more than 3 times of the normal upper limit, total bilirubin (TBIL) more than 2 times of the normal upper limit;
9. Creatinine levels ≥ 1.4 mg/dL (123μmol/L) or creatinine clearance ≤ 50 ml/min;
10. History of malignant tumors;
11. Simultaneous participation in another clinical study with investigational medicinal product(s) or researcher thinks the subjects are not suitable for this trial.

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1160 (Estimated)
Dates: Start 2018-09-15 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of uterine fibroids in different groups | two years after treatment
  Incidence rate of uterine fibroids in different groups after two years treatment

SECONDARY OUTCOMES:
Hypercalcemia | Two years after treatment
  The level of serum calcium > 2.5 mmol/L
abnormal liver function | Two years after treatment
  Alanine aminotransferase (ALT) or aspartate transaminase (AST) more than 3 times of the normal upper limit, or total bilirubin (TBIL) more than 2 times of the normal upper limit
abnormal renal function | Two years after treatment
  Creatinine levels≥1.4 mg/dL (123μmol/L) or creatinine clearance ≤ 50 mL/min
Incidence rate of uterine fibroids in different groups | One year after treatment
  Incidence rate of uterine fibroids in different groups after one year treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Sheng B, Song Y, Liu Y, Jiang C, Zhu X. Association between vitamin D and uterine fibroids: a study protocol of an open-label, randomised controlled trial. BMJ Open. 2020 Nov 6;10(11):e038709. doi: 10.1136/bmjopen-2020-038709. PMID 33158822

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT03586947/Prot_SAP_000.pdf